CLINICAL TRIAL: NCT04514289
Title: Endometrium Kanseri Nedeniyle Opere Olacak hastaların Sentinel Lenf Nodu Diseksiyonu değerlendirilirken kullanılan Iki farklı yöntemin kıyaslaması
Brief Title: To Assess and Compare the Performance Two Approach for Sentinel Lymph Node (SNLD) Biopsy for Endometrial Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Haseki Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Cihan Comba, gynecological oncology specialist, Haseki Training and Research Hospital
Other Study IDs: 20-2020
Record Dates: First submitted 2020-07-29; First posted 2020-08-14 (Actual); Last update posted 2020-08-14 (Actual); Status verified 2020-08

CONDITIONS: Endometrial Cancer; Sentinel Lymph Node; Indocyanine Green
MeSH Terms: conditions — Endometrial Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- assesment SLND with enjection by using ICG: Patients who have endometrium cancer; undergo sentinel lymph node detection by using fluorescence imaging with an indocyanine green solution. Two different ways used to assess SLND. The first group in which the cervix is injected superficially with 1 mL of ICG ( indocyanine green) at 4 and 8 o'clock quadrans.
  Interventions: Drug: Indocyanine green solution
- assesment SLND with hysterescopy by using ICG: Patients who have endometrium cancer; undergo sentinel lymph node detection by using fluorescence imaging with an indocyanine green solution. Two different ways used to assess SLND. The second one which ICG has injected the uterine cavity during hysteroscopy. Our aim is to assess and compare the performance two approaches for sentinel lymph node ( SLND) biopsy.
  Interventions: Drug: Indocyanine green solution

INTERVENTIONS:
Drug: Indocyanine green solution — Indocyanine green (ICG) is a cyanine dye used in medical diagnostics.ICG is a fluorescent dye that is used in medicine as an indicator substance.
  Other Names: No indocyanine green solution

SUMMARY:
to assess and compare the performance two approaches for sentinel lymph node ( SLND) biopsy

DETAILED DESCRIPTION:
Endometrial cancer is the most common gynecologic cancer. Most patients diagnosed in early stages because cancer causes remarkable symptoms such as postmenopausal or abnormal bleeding. Mostly, it does not spread, detects no metastasis. Endometrial carcinoma is surgically staged. Laparotomy or minimally invasive surgery can be performed for treatment and staging. Patients have been operated for staging surgery, have a larger surgical incision, longer operation period, more complications, more intensive care units need. Nowadays, researchers show us that there is no difference in overall survival and prognosis between surgery with or without lymphadenectomy in endometrial cancer. With all these improvements in gynecologic oncology leads us to minimally invasive surgery. Patients undergo sentinel lymph node detection by using fluorescence imaging with an indocyanine green solution. Two different ways used to assess SLND. The first group who the cervix is injected superficially with 1 mL of ICG ( indocyanine green) at 4 and 8 o'clock quadrans. The second group who ICG has injected the uterine cavity during hysteroscopy. The investigator's aim is to assess and compare the performance of two approaches for sentinel lymph node ( SLND) biopsy.

ELIGIBILITY:
Inclusion Criteria:

* The patient must be willing and able to provide informed consent
* The patient is willing and able to comply with the study protocol
* The patient has endometrial cancer and is performed SLND
* The patient agrees to follow-up examination out to 5-years post-treatment

Exclusion Criteria:

* The patient is not a candidate for surgery
* The patient has metastasis
* The patient has known or suspected allergies to iodine, indocyanine green( ICG)

Ages: 18 Years to 90 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female
Study Population: patients who have experienced endometrial cancer surgery
Sampling Method: Non-Probability Sample
Enrollment: 106 (Estimated)
Dates: Start 2020-03-01 (Actual); Primary Completion 2021-06-30 (Estimated); Study Completion 2021-08-30 (Estimated)

PRIMARY OUTCOMES:
SLN detecting rate | 1 year
  SLN is the first lymph node to spread tumoral cells.

SECONDARY OUTCOMES:
Overall survival | 5 years
  Overall survival of endometrial cancer measures as five years
Disease free survival | 5 years
  Disease free survival can be describe with no tumor occurance after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Cihan Comba, M.D., Study Chair — Sultangazi Haseki Training and Research Hospital
Locations (1):
- Cihan Comba, Istanbul, Sultangazi, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided